CLINICAL TRIAL: NCT01997645
Title: Ligation of Intersphincteric Fistula Tract (LIFT) Versus Rectal Advanced Mucosal Flap (RAF) in Surgical Treatment of High Perianal Fistulas
Brief Title: Surgical Treatment of High Perianal Fistulas
Acronym: LIFTRAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Otakar Sotona, MD, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FN HK CP 2013
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Anal Fistula; Rectal Fistula
Keywords: Anal fistula; Rectal fistula; Intersphincteric fistula; Perianal fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rectal advanced mucosal flap (Active Comparator): Procedure will be performed in general anesthesia without mechanical bowel preparation. Antibiotic prophylaxis (Metronidazole 1g) will be applied intravenously 60 minutes prior the surgery.
  In RAF procedure, internal opening will identified and after infiltration with saline-adrenalin solution (1/100000) the mucosal flap will be mobilized proximally. The external tract and internal opening will be excised and the defect will be sutured. After that, the flap will be advanced from both sides with absorbable suture and overlapped over the internal opening. External openings will be left open.
  Interventions: Procedure: RAF
- Ligation of intersphincteric fistula tract (Active Comparator): Procedure will be performed in general anesthesia without mechanical bowel preparation. Antibiotic prophylaxis (Metronidazole 1g) will be applied intravenously 60 minutes prior the surgery.
  Before LIFT procedure the fistula tract will be identified with small probe. The intersphincteric space will be reached by dissection from small (2-4cm) incision. The fistula tract will be divided and ligated on both sides with Polydioxanone (PDS) suture. The external and internal openings will be left open to drain.
  Interventions: Procedure: LIFT

INTERVENTIONS:
Procedure: LIFT
  Arms: Ligation of intersphincteric fistula tract
Procedure: RAF
  Arms: Rectal advanced mucosal flap

SUMMARY:
Perianal fistula is a chronic phase of anorectal infection that occurs predominantly in the third and fourth decade of life. According to Parks classification fistulas have been divided into intersphincteric, transsphincteric, suprasphincteric and extrasphincteric. Simple fistulotomy can be performed with satisfactory outcomes in low fistula tracts but in high (transsphincteric) fistulas it may affect anal continence seriously.

Therefore sphincter preserving procedures should be preferred in these cases. Rectal advancement mucosal flap (RAF) is one of the methods used in surgical fistula eradication with high success rate in cryptoglandular fistulas. However, this technique is technically demanding and results can be expert depended with wide spread of healing rates (24-100%) in individual studies as referred in recent systematic review.

Ligation of the intersphincteric fistula tract (LIFT) has been presented in 2007 as a simple sphincter preserving technique. The success rate varies between 40-95% with low overall incontinence rate (6%).

The aim of the study is to compare the efficacy of the LIFT and RAF procedure for treatment of high perianal fistulas.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or older
* Diagnosis of simple intersphincteric or transsphincteric fistula
* Patients able to comply with the study protocol as per investigator criteria
* Signed and dated informed consent by the patient
* Absence of any exclusion criteria

Exclusion Criteria:

* Recurrent anal fistula
* Suprasphincteric, low subcutaneous fistula
* Multiple fistulas
* Posttraumatic fistula
* Perianal hidradenitis
* Fistula arises from other than cryptoglandular origin
* Previous anal surgery except of abscess
* Inflammatory Bowel Disease
* History of fecal incontinence
* Rectal prolapse
* Malignant disease and life expectancy of less than 1 year, or chemotherapy and radiotherapy less than six months prior enrolment
* HIV infection
* Pregnancy
* Participation in another clinical trial less than one month prior to enrolment, or involvement in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | One year
  Fistula recurrence will be defined according to AGA (American Gastroenterological Association) criteria as a purulent secretion from external fistula opening followed the compression.
  Fistula recurrence will be confirmed by evaluation under anesthesia (followed by drainage).

SECONDARY OUTCOMES:
Postoperative pain | 14 days
  Postoperative pain will be assessed 4 times per day during the first 2 postoperative days (VAS - visual analogue scale), after that 3 times per day over next 14 days (patient's diary).
Pre- and postoperative continence | One year
  Pre- and postoperative continence will be evaluated with Wexner score.
Postoperative morbidity | One month
  Will be evaluated according to Clavien-Dindo classification.
Quality of life | One year
  For quality of life evaluation SF-36 questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Július Örhalmi, MD, Principal Investigator — University Hospital Hradec Kralove; Zuzana Šerclová, MD, Principal Investigator — Central MIlitary Hospital Prague; Karel Klos, MD, Principal Investigator — District Hospital Nový Jičín
Locations (3):
- Czechia (3):
  - Department of Surgery, Charles University, Faculty of Medicine and University Hospital, Hradec Králové
  - Departement of Surgery, District Hospital, Nový Jičín
  - Departement of Surgery, Military University Hospital, Prague

REFERENCES:
- [Background] Marks CG, Ritchie JK. Anal fistulas at St Mark's Hospital. Br J Surg. 1977 Feb;64(2):84-91. doi: 10.1002/bjs.1800640203. PMID 890252
- [Background] Parks AG, Gordon PH, Hardcastle JD. A classification of fistula-in-ano. Br J Surg. 1976 Jan;63(1):1-12. doi: 10.1002/bjs.1800630102. PMID 1267867
- [Background] Malik AI, Nelson RL. Surgical management of anal fistulae: a systematic review. Colorectal Dis. 2008 Jun;10(5):420-30. doi: 10.1111/j.1463-1318.2008.01483.x. PMID 18479308
- [Background] Garcia-Aguilar J, Belmonte C, Wong DW, Goldberg SM, Madoff RD. Cutting seton versus two-stage seton fistulotomy in the surgical management of high anal fistula. Br J Surg. 1998 Feb;85(2):243-5. doi: 10.1046/j.1365-2168.1998.02877.x. PMID 9501826
- [Background] Soltani A, Kaiser AM. Endorectal advancement flap for cryptoglandular or Crohn's fistula-in-ano. Dis Colon Rectum. 2010 Apr;53(4):486-95. doi: 10.1007/DCR.0b013e3181ce8b01. PMID 20305451
- [Background] Rojanasakul A, Pattanaarun J, Sahakitrungruang C, Tantiphlachiva K. Total anal sphincter saving technique for fistula-in-ano; the ligation of intersphincteric fistula tract. J Med Assoc Thai. 2007 Mar;90(3):581-6. PMID 17427539
- [Background] Yassin NA, Hammond TM, Lunniss PJ, Phillips RK. Ligation of the intersphincteric fistula tract in the management of anal fistula. A systematic review. Colorectal Dis. 2013 May;15(5):527-35. doi: 10.1111/codi.12224. PMID 23551996
- [Background] Sandborn WJ, Fazio VW, Feagan BG, Hanauer SB; American Gastroenterological Association Clinical Practice Committee. AGA technical review on perianal Crohn's disease. Gastroenterology. 2003 Nov;125(5):1508-30. doi: 10.1016/j.gastro.2003.08.025. No abstract available. PMID 14598268
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542